CLINICAL TRIAL: NCT03657654
Title: Voice Outcomes Following Thyroidectomy Compared to Surgeries That Do Not Involve Risk to the Laryngeal Nerves
Brief Title: Voice Outcomes Following Thyroidectomy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, David Shonka, MD, Associate Professor, University of Virginia
Other Study IDs: 20892
Record Dates: First submitted 2018-08-29; First posted 2018-09-05 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Thyroid Cancer; Thyroid Nodule
Keywords: Thyroidectomy; Laryngeal Nerves; Voice problems
MeSH Terms: conditions — Thyroid Neoplasms; Thyroid Nodule

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Thyroidectomy: Patients that are clinically referred for a thyroidectomy for known or potential cancer.
  Interventions: Other: No intervention: observational only
- Other surgeries: Patients must be clinically referred for a surgery requiring intubation, but without risk to the laryngeal nerves or dissection adjacent to the larynx
  Interventions: Other: No intervention: observational only

INTERVENTIONS:
Other: No intervention: observational only — No intervention: observational only

SUMMARY:
This is an observational study of voice outcomes in participants following thyroidectomy or another head and neck surgery that does not involve risk to the larynx other than risks incurred due to intubation alone. These comparative (non-thyroidectomy) surgeries would not be expected to interfere with the primary nerves involved with voice production, so they would help to better understand the effect of intubation alone on voice outcomes.

DETAILED DESCRIPTION:
Voice difficulty is a common complaint following thyroidectomy, and while the procedure risks injury to laryngeal nerves involved in voice production, voice difficulty is common even in the absence of evident injury to these nerves. The cause of voice change in these situations is not well defined, and multiple mechanisms have been suggested. Some potential mechanisms include trauma to the laryngeal skeleton from intraoperative manipulation of the strap muscles, cricothyroid muscle, thyroid, cartilage, or trachea. However, it is also possible that irritation due to intubation and edema to the neck and oral or pharyngeal soft tissues that develops after the surgery as a result of intubation plays a role in postoperative voice change. These mechanisms can occur in any operation requiring general endotracheal anesthesia even when the laryngeal nerves are not specifically at risk of injury.

The purpose of this study is to evaluate voice outcomes after thyroidectomy (both objective and subjective patient and clinician reported) and compare those to voice outcomes after other surgeries that do not put the recurrent or superior laryngeal nerves at risk or traumatize the laryngeal skeleton, but do require general endotracheal anesthesia. The primary assessment tool will be the Voice Handicap Index-10 (VHI-10), which is a questionnaire that asks about the patient's interpretation of his/her voice quality and the impact it is having on daily activities. Data analysis will be done to see if participants have a significant change in their pre-operation VHI-10 score at approximately 1 week and 3 months post-operation. Additional assessments tools will include nasolaryngoscopy and nasolaryngeal stroboscopy to assess global vocal fold function, Consensus Auditory Perceptual Evaluation of Voice (CAPE-V) and computerized speech lab (CSL) acoustics to assess voice quality, and vocal aerodynamic analysis to determine air flow through the larynx.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Age ≥ 18 years
4. Subject must be clinically referred for a thyroidectomy for known or potential cancer, or subject must be clinically referred for a surgery requiring intubation, but without risk to the laryngeal nerves or dissection adjacent to the larynx for the control group
5. As the VHI-10 is not available and validated in all languages, participants must be able to comprehend a validated version of the VHI-10 in their language

Exclusion Criteria:

1. Plan to include neck dissection in upcoming surgery (control group/non-thyroidectomy patients only)
2. Known to be pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults that have been clinically referred for thyroidectomy or another surgery requiring intubation but without risk to the laryngeal nerves or dissection adjacent to the larynx.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2019-04-23 (Actual); Primary Completion 2023-12-15 (Estimated); Study Completion 2023-12-15 (Estimated)

PRIMARY OUTCOMES:
Change in Voice Handicap Index-10 (VHI-10) score before and after surgery | Baseline, 1 week following surgery, 3 months following surgery
  This is a VHI-10 is a questionnaire that asks about the patient's interpretation of his/her voice quality and the impact it is having on daily activities.

SECONDARY OUTCOMES:
Video flexible nasolaryngoscopy | Within 24 hours following surgery
  This procedure is endoscopic and allows for visualization and audio/video recording of the vocal folds at rest and during speech
Video nasolaryngeal stroboscopy | Baseline, 1 week following surgery, 3 months following surgery
  This imaging is another form of nasolaryngoscopy but has the addition of a strobe light. The strobe light provides an optical illusion in which the vocal cords appear to be moving in slow motion on the video, even though its movement is unaltered.
Vocal Aerodynamics Analysis | Baseline, 1 week following surgery, 3 months following surgery
  This assessment is performed by fitting the participant with a mask that is attached to a tube that goes just inside the participant's lips. This positioning allows for the participant to close his/her lips around the tube without occluding it. The participant is asked to produce repeated syllables like pi-pi-pi-pi-pi, which allows for airflow and air pressure to be measured and reflects vocal fold function.
CAPE-V | Baseline, 1 week following surgery, 3 months following surgery
  The CAPE-V is a tool used for clinical auditory-perceptual assessment of voice. It is intended to describe the severity of various auditory attributes of a voice problem, and it is determined by the clinician's auditory assessment of the patient's voice.
CSL acoustics | Baseline, 1 week following surgery, 3 months following surgery
  This assessment involves having the participant speak into a microphone. The patient says a few scripted sentences, as well as repeated sounds, which is then analyzed by the computer software. The assessment allows for determination of vocal loudness, pitch, and voice quality. Voice quality is determined based on measures including vocal shimmer, vocal jitter, and background noise in the voice. Shimmer measures variation in voice amplitude and jitter measures variation in frequency.

CONTACTS AND LOCATIONS:
Overall Officials: David C Shonka, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No